CLINICAL TRIAL: NCT06608511
Title: Liquid Biomarker Study in Melanoma and Non-Melanoma Skin Cancers
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2024-1143; KL2TR002374-07 (NIH); UW24066 (Other: UW Madison); A534260 (Other: UW Madison); Protocol Version 9/9/24 (Other: UW Madison)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Skin Cancer; Melanoma (Skin Cancer); Basal Cell Carcinoma of Skin; Basal Cell Carcinoma of Skin, Site Unspecified; Cutaneous Squamous Cell Carcinoma (CSCC); Merkel Cell Carcinoma of Skin
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Basal Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Skin cancer: Participants with melanoma or non-melanoma skin cancer
  Interventions: Other: Blood draw for the laboratory assessment

INTERVENTIONS:
Other: Blood draw for the laboratory assessment — Participants will have 50 milliliters (3.5 tablespoons) of blood drawn

SUMMARY:
The goal of this observational study is to study blood samples and compare them to other biospecimens and clinical outcomes in participants who have melanoma or non-melanoma skin cancers. The main question it aims to answer is:

* Are blood based signatures able to predict progression-free survival (PFS)?

Participants undergoing regular treatment for their skin cancer will provide blood samples.

DETAILED DESCRIPTION:
This observational study is being done to identify possible biomarkers that can be used for prognostic, prediction, or monitoring considerations in patients with melanoma or non-melanoma skin cancer undergoing treatment. Investigators plan to investigate blood factors which include circulating tumor cells (CTCs - i.e., cancer cells that can be detected in the blood) and their associated protein and mRNA expression; circulating tumor DNA (ctDNA - i.e., pieces of DNA from cancer cells that can be found in the blood); and tumor-derived exosomes (i.e., extracellular vesicles generated by cancer cells that carry nucleic acids, proteins, and metabolites).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Participants must meet at least one of the following criteria:
* Finding suspicious of melanoma or non-melanoma skin cancer based on clinical, radiographic, or laboratory findings. Non-melanoma skin cancers include: basal cell carcinoma, cutaneous squamous cell carcinoma, and Merkel cell carcinoma.
* A confirmed diagnosis of melanoma or non-melanoma skin cancer.

Exclusion Criteria:

* Vulnerable populations, including pregnant women, those who lack consent capacity, the mentally ill, prisoners, cognitively impaired persons, children (age <18), and UW employees that report to the investigator(s) or to study team members.
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be from the Melanoma Medical Oncology Clinic at the Carbone Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in tumor-derived exosomes and progression free survival | Baseline to progression, up to 3 years
  To investigate whether changes in tumor-derived exomes measured in serum could represent a potential prognostic biomarker, measured as progression free survival (the duration of time from Day 1 of treatment to time of progression based on clinical or radiographic grounds) or death as a results of any cause, whichever occurs first.
Change in circulating tumor cells and progression free survival | Baseline to progression, up to 3 years
  To investigate whether changes in circulating tumor cells measured in serum could represent a potential prognostic biomarker, measured as progression free survival (PFS). PFS is the duration of time from Day 1 of treatment to time of progression (based on clinical or radiographic grounds) or death as a result of any cause, whichever occurs first.
Change in circulating tumor DNA and progression free survival | Baseline to progression, up to 3 years
  To investigate whether changes in circulating tumor DNA measured in serum could represent a potential prognostic biomarker, measured as progression free survival. PFS is the duration of time from Day 1 of treatment to time of progression (based on clinical or radiographic grounds) or death as a result of any cause, whichever occurs first
Change in tumor-derived exosomes and overall survival | Baseline to progression, up to 3 years
  To investigate whether changes in tumor-derived exomes measured in serum could represent a potential prognostic biomarker measured as overall survival (OS). OS - the duration of time from Day 1 of treatment to time of death as a result of any cause.
Change in circulating tumor cells and overall survival | Baseline to progression, up to 3 years
  To investigate whether changes in circulating tumor cells measured in serum could represent a potential prognostic biomarker measured as overall survival. OS - the duration of time from Day 1 of treatment to time of death as a result of any cause.
Change in circulating tumor DNA and overall survival | Baseline to progression, up to 3 years
  To investigate whether changes in circulating tumor DNA measured in serum could represent a potential prognostic biomarker measured as overall survival. OS - the duration of time from Day 1 of treatment to time of death as a result of any cause
Change in tumor-derived exosomes and treatment response | Baseline to progression, up to 3 years
  To investigate whether changes in tumor-derived exomes measured in serum could represent a potential prognostic biomarker measured as treatment response. Treatment response - rate of objective response (partial response + complete response) and disease control rate (stable disease + partial response + complete response) per RECIST v1.1
Change in circulating tumor cells and treatment response | Baseline to progression, up to 3 years
  To investigate whether changes in circulating tumor cells measured in serum could represent a potential prognostic biomarker measured as response to treatment. Treatment response - rate of objective response (partial response + complete response) and disease control rate (stable disease + partial response + complete response) per RECIST v1.1
Change in circulating tumor DNA and treatment response | Baseline to progression, up to 3 years
  To investigate whether changes in circulating tumor DNA measured in serum could represent a potential prognostic biomarker measured as response to treatment. Treatment response - rate of objective response (partial response + complete response) and disease control rate (stable disease + partial response + complete response) per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ma, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No